CLINICAL TRIAL: NCT00547066
Title: A Phase I/II Study of Immunotherapy With Humanized Anti-CD20 Antibody, IMMU-106 (hA20), in Adult Patients With Chronic Immune Thrombocytopenic Purpura
Brief Title: Study of Veltuzumab (hA20) at Different Doses in Patients With ITP
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hA20-07
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2020-03

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Autoimmune Thrombocytopenic Purpura; Purpura, Thrombocytopenic, Autoimmune
Keywords: ITP; hA20; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — veltuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- veltuzumab (Experimental): veltuzumab is a humanized CD20 antibody administered subcutaneously.
  Interventions: Biological: veltuzumab

INTERVENTIONS:
Biological: veltuzumab — hA20 will be administered intravenously in two doses over two weeks
  Other Names: IMMU-106; hA20; humanized anti-CD20

SUMMARY:
This trial will study different dose levels of hA20 (IMMU-106) to see if they are safe and effective for treating ITP.

DETAILED DESCRIPTION:
The goal of current treatment guidelines for most patients with chronic adult ITP is to maintain platelet levels above 30 x 109/L. The conventional first-line therapy is corticosteroids with or without intravenous immunoglobulins, but many patients relapse when steroids are tapered. Standard therapy then is splenectomy, but patients with refractory ITP who do not respond require further therapy. Unfortunately, immunosuppressive agents or other available treatments typically produce only short-term responses. Because of the lack of medical options after first-line therapy, the target population for this first study of anti-CD20 immunotherapy with hA20 are adult patients with chronic ITP who failed at least one standard ITP therapy (i.e., received at least one standard ITP therapy and now present with platelet levels below 30 x 109/L).

In autoimmune disease, rituximab as well as other anti-CD20 antibodies currently being considered for commercialization have focused on a different dosing schedule in rheumatoid arthritis, and use fixed dosages rather than variable doses based on body surface area. In addition, recent studies of these newer anti-CD20 antibodies in rheumatoid arthritis have reported that lower doses indeed appear effective when administered twice, 2 weeks apart. Based upon these considerations, patients in this study will receive hA20 twice, 2 weeks apart, and administered at one of 3 dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years old, with or without prior splenectomy
* Signed written informed consent obtained prior to study entry
* ITP according to ASH guidelines, with other potential causes of thrombocytopenia excluded
* Platelet levels < 150 x 109/L for more than 6 months
* Received an adequate course of at least one standard ITP treatment (an inadequate course of standard ITP therapy does not qualify as meeting this requirement)
* Platelet count < 30 x 109/L at study entry and on at least one other occasion at least 1 week apart within the past month. (Phase I only: platelet count also > 10 x 109/L at study entry).
* Bleeding assessment score of Grade 0 or 1. See full protocol for all inclusion criteria

Exclusion Criteria:

See full protocol for exclusion criteria or contact study staff for details

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Primary - Safety | 1 year
  Hematology laboratory results and adverse events will be followed closely for one year.
Secondary - Efficacy | 5 years
  Platelet responses will be followed for up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PHD, Study Chair — Gilead Sciences
Locations (8):
- United States (8):
  - University of Southern California- Keck School of Medicine, Los Angeles, California
  - Center of Hope for Cancer and Blood Disorders, Riverdale, Georgia
  - Georgia Cancer Specialtists, Tucker, Georgia
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Hematology Oncology Specialists, Metairie, Louisiana
  - Denville, New Jersey
  - Hematology/Oncology Specialists, Buffalo, New York
  - New York Presbyterian Hospital Weill Cornell Medical Center, New York, New York

REFERENCES:
- [Derived] Liebman HA, Saleh MN, Bussel JB, Negrea OG, Horne H, Wegener WA, Goldenberg DM. Comparison of two dosing schedules for subcutaneous injections of low-dose anti-CD20 veltuzumab in relapsed immune thrombocytopenia. Haematologica. 2016 Nov;101(11):1327-1332. doi: 10.3324/haematol.2016.146738. Epub 2016 Aug 11. PMID 27515248
- [Derived] Liebman HA, Saleh MN, Bussel JB, Negrea OG, Horne H, Wegener WA, Goldenberg DM. Low-dose anti-CD20 veltuzumab given intravenously or subcutaneously is active in relapsed immune thrombocytopenia: a phase I study. Br J Haematol. 2013 Sep;162(5):693-701. doi: 10.1111/bjh.12448. Epub 2013 Jul 6. PMID 23829485